CLINICAL TRIAL: NCT05458518
Title: A Randomised Controlled Trial on the Timing of Wound Dressing Removal After Emergency Caesarean Delivery
Brief Title: Caesarean Wound Dressing Removal Study
Acronym: Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Kemaman (Other)
Responsible Party: Principal Investigator, Zahar Azuar Zakaria, Consultant, Head of Department, Lead Investigator, Hospital Kemaman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMRR ID-22-00321-NZM
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Surgical Wound; Surgical Wound Infection; Cesarean Section Complications
Keywords: wound dressing; cesarean
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dressing removal at 24 hours (Active Comparator): The wound dressing will be removed 24 hours after emergency cesarean delivery
  Interventions: Procedure: Cesarean wound dressing removal
- Dressing removal at 48 hours (Placebo Comparator): The wound dressing will be removed 48 hours after emergency cesarean delivery
  Interventions: Procedure: Cesarean wound dressing removal

INTERVENTIONS:
Procedure: Cesarean wound dressing removal — The cesarean wound dressing is to be removed and the surgical wound exposed

SUMMARY:
An open labelled randomised trial on the timing of wound dressing removal for emergency caesarean delivery in labour.

DETAILED DESCRIPTION:
The trial is unblinded randomised trial on surgical wound dressing at 24 versus 48 hours after the emergency caesarean delivery in labour.

The primary outcome is the prevalence of wound complications (hematoma, seroma, infection/ dehiscence) The secondary objectives are the maximum pain after the surgery (in ward) and the timing of the patient's first bath after the surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Lower segment caesarean delivery
3. Primary or repeat caesarean delivery
4. Caesarean section in active phase of labour.
5. Regional anaesthesia

Exclusion Criteria:

1. Upper segment or classical caesarean delivery
2. Massive postpartum haemorrhage > 1.5 litre
3. Pre-delivery chorioamnionitis
4. Skin closure using interrupted suture
5. Acquired or congenital coagulation disorder
6. Associated medical or obstetric condition requiring prolonged hospital stay after delivery such as severe pre-eclampsia, uncontrolled diabetes mellitus, cardiac disease, systemic infection.
7. Inability to give consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cesarean wound complication | 30 days
  Hematoma, seroma, wound infection, wound dehiscence

SECONDARY OUTCOMES:
Pain control | 48 hours
  Perceived pain after caesarean according to Visual Analogue Scale (0/10 = no pain; 10/10 = worst pain)
Self hygiene | 48 hours
  Timing of first bath after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zahar A Zakaria, MD, Principal Investigator — Hospital Kemaman
Locations (1):
- Hospital Kemaman, Kampong Kemaman, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peleg D, Eberstark E, Warsof SL, Cohen N, Ben Shachar I. Early wound dressing removal after scheduled cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol. 2016 Sep;215(3):388.e1-5. doi: 10.1016/j.ajog.2016.03.035. Epub 2016 Mar 25. PMID 27018465
- [Result] Kilic GS, Demirdag E, Findik MF, Tapisiz OL, Sak ME, Altinboga O, Sak S, Unlu BS, Evsen MS, Zeybek B, Borahay M, Kuo YF. Impact of timing on wound dressing removal after caesarean delivery: a multicentre, randomised controlled trial. J Obstet Gynaecol. 2021 Apr;41(3):348-352. doi: 10.1080/01443615.2020.1736015. Epub 2020 Apr 21. PMID 32312139
- [Result] Tan PC, Rohani E, Lim M, Win ST, Omar SZ. A randomised trial of caesarean wound coverage: exposed versus dressed. BJOG. 2020 Sep;127(10):1250-1258. doi: 10.1111/1471-0528.16228. Epub 2020 Apr 16. PMID 32202035
- [Result] Zhang T, Zhang F, Chen Z, Cheng X. Comparison of early and delayed removal of dressing following primary closure of clean and contaminated surgical wounds: A systematic review and meta-analysis of randomized controlled trials. Exp Ther Med. 2020 May;19(5):3219-3226. doi: 10.3892/etm.2020.8591. Epub 2020 Mar 11. PMID 32266018